CLINICAL TRIAL: NCT05562063
Title: SOTA-P-CARDIA Trial: A Randomized Trial of Sotagliflozin in HFpEF Patients Without Diabetes
Brief Title: Sotagliflozin in Heart Failure With Preserved Ejection Fraction (HFpEF) Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Juan Badimon (Other)
Responsible Party: Sponsor-Investigator, Juan Badimon, Professor of Medicine, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GCO-22-0574
Record Dates: First submitted 2022-09-27; First posted 2022-09-30 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Heart Failure With Preserved Ejection Fraction
MeSH Terms: interventions — (2S,3R,4R,5S,6R)-2-(4-chloro-3-(4-ethoxybenzyl)phenyl)-6-(methylthio)tetrahydro-2H-pyran-3,4,5-triol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sotagliflozin (Experimental): Daily administration of sotagliflozin (2x200 mg, orally, once a day) for 6 months.
  Interventions: Drug: Sotagliflozin
- Placebo (Placebo Comparator): Daily administration of placebo (2 tablet identical in appearance and color to sotagliflozin tablets, orally, once a day) for 6 months.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sotagliflozin — Daily administration of sotagliflozin (2x200 mg, PO, OD) for 6 months.
  Arms: Sotagliflozin
Drug: Placebo — Matching placebo for 6 months.
  Arms: Placebo

SUMMARY:
The clinical benefits of the dual Sodium-Glucose cotransporter (SGLT) 1 and 2-inhibition have recently been reported in two clinical trials. The SOLOIST reported the benefits of sotagliflozin in Type-2 Diabetes Mellitus (T2DM) patients hospitalized for worsening of Heart Failure (HF), while the SCORED involved T2DM patients with Chronic Kidney Disease (CKD). It is worth noting that not only did the event curves separate within the first week post-treatment, but the effects of sotagliflozin on HF-related outcomes were observed regardless of Left Ventricular Ejection Fraction (LVEF) values and did not seem to attenuate with increasing LVEF as seen with empagliflozin and sacubitril/valsartan. Despite the favorable outcomes, the mechanism(s) of action through which sotagliflozin exerts these benefits remains unclear.

The present study aims to investigate the potential (non-glucose dependent) "cardio-renal" pleiotropic effects of sotagliflozin in a mechanistic, randomized, double blind, placebo-control trial in HF patients with preserved ejection fraction (HFpEF). Comparisons between treatment groups will be made using cardiac MRI, CPET, 6-MWT and KCCQ-12.

ELIGIBILITY:
Inclusion Criteria: patients should meet all of the following criteria

* Ambulatory patients age ≥ 18 years
* Written informed consent prior to admission to the trial.
* No diabetes as confirmed by HbA1c <6.5%, fasting serum glucose <126 mg/dL, and review of concomitant medications and medical history
* Diagnosis of Heart failure (NYHA II to III)
* LVEF > 50%
* On medical therapy for heart failure consistent with prevailing cardiovascular guidelines at a stable dose for ≥4 weeks prior to screening, except for diuretics which must have been stable for ≥2 weeks prior to screening
* Women of child-bearing potential must agree to use birth control measures with a failure rate of <1% per year during the treatment period of the study

Exclusion Criteria:

* Type 1 and Type 2 diabetes
* Acute coronary syndrome (ACS) or cardiac surgery within the last week.
* Pregnant or lactating women,
* Acute decompensated HF or hospitalized for HF within 1 month from screening visit
* Glomerular Filtration Rate (GFR) < 25 ml/ min/1.73m2,
* Patients on drugs with potential interaction with sotagliflozin including digoxin, phenytoin, HIV medication and rifampin.
* Receiving SGLT2-I 3-months prior to randomization.
* non-MRI compatible PM or ICD and any other medical or physical condition considered unappropriated by a study physician.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2022-10-26 (Actual); Primary Completion 2025-06-04 (Actual); Study Completion 2025-06-04 (Actual)

PRIMARY OUTCOMES:
Changes in Left Ventricular mass in CMRI | Baseline and 6 months
  Changes in Left Ventricular (LV) mass at 6 months compared to baseline

SECONDARY OUTCOMES:
Changes in Left Ventricular end-systolic volume | Baseline and 6 months
  Changes in left ventricular end-systolic volume (LVESV) in CMRI at 6 months compared to baseline
Changes in Left Ventricular end-diastolic volume | Baseline and 6 months
  Changes in left ventricular end-diastolic volume (LVEDV) in CMRI at 6 months compared to baseline
Changes in extracellular volume (ECV) | Baseline and 6 months
  Changes in extracellular volume (ECV) to assess Left Ventricular interstitial myocardial fibrosis as quantified using T1 mapping at 6 months compared to baseline
Changes in Left atrial volume index | Baseline and 6 months
  Changes in Left atrial volume index measured by CMRI at 6 months compared to baseline
Changes in Peak oxygen consumption (peakVO2) | Baseline and 6 months
  Changes in exercise capacity as assessed by peak oxygen consumption in Cardiopulmonary exercise test (CPET) at 6 months compared to baseline
Changes 6 minute walk test | Baseline and 6 months
  Changes in exercise tolerance as assessed by 6 minute walk test, or the distance covered over a time of 6 minutes, at 6 months compared to baseline
Changes in The Kansas City Cardiomyopathy Questionnaire (KCCQ) | Baseline and 6 months
  Changes in The KCCQ at 6 months compared to baseline. The KCCQ is the most widely used instrument to evaluate quality of life in Heart Failure (HF).
  The KCCQ is a 12-item self-administered questionnaire used to measure the patient's perception of their health status. The KCCQ is a disease-specific health status instrument composed of 12 items that quantifies the domains of physical limitations, symptoms, self-efficacy, social limitation and quality of life from heart failure. Full scale range is from 0 to 100; higher scores reflect better health status.

CONTACTS AND LOCATIONS:
Overall Officials: Juan J Badimon, Principal Investigator — Icahn School of Medicine at Mount Sinai; Carlos G Santos-Gallego, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Undecided: It is not yet known if there will be a plan to make IPD available.